CLINICAL TRIAL: NCT05407597
Title: Prospective, Randomised, Double-blind Trial of Icatibant Compared to Placebo in Patients With Early Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) Infection
Brief Title: Inhibition of Bradykinin in COVID-19 Infection With Icatibant
Acronym: ICASARS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21036JK-AS; 2021-005851-35 (EudraCT Number)
Record Dates: First submitted 2022-05-11; First posted 2022-06-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: SARS CoV 2 Infection
Keywords: Bradykinin; Alveolar-arterial gradient; Interleukin-6 (IL-6)
MeSH Terms: conditions — COVID-19 | interventions — icatibant; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either Icatibant (30mg) or 0.9% Sodium Chloride (3mls)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and investigators will be blinded to treatment allocation. An unblinded research nurse will administer the study medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Icatibant and Standard of care (SOC) (Active Comparator): Icatibant will be given as a single, subcutaneous injection
  Interventions: Drug: Icatibant
- 0.9% Sodium Chloride and Standard of care (SOC) (Placebo Comparator): Placebo will be given as a single, subcutaneous injection
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Icatibant — Solution for injection, 30mg (3mls) administered as a single subcutaneous injection
  SARS CoV-2 patients will receive all supportive treatment and medications that are used as standard of care including but not limited to Dexamethasone, Remdesivir, Tocilizumab and antibiotics.
  Arms: Icatibant and Standard of care (SOC)
Drug: 0.9% Sodium Chloride Injection — Solution for injection (3mls) administered as a single subcutaneous injection
  SARS CoV-2 patients will receive all supportive treatment and medications that are used as standard of care including but not limited to Dexamethasone, Remdesivir, Tocilizumab and antibiotics.
  Arms: 0.9% Sodium Chloride and Standard of care (SOC)

SUMMARY:
There is excess accumulation of bradykinin during symptomatic SARS CoV-2 lung infection. Bradykinin causes oedema in the lung, with reduced oxygen. It also causes vasodilation, hypotension and cytokine release.

DETAILED DESCRIPTION:
In a normal reaction to a wound, such as after surgery, there is stimulation of pain nerves (called c-fibres), swelling and clotting. When people are hospitalized with COVID-19 they usually have a cough (lung c-fibre stimulation), swelling in the lung and clotting.

Bradykinin is a chemical that is released in response to inflammation. It causes C-fibre stimulation, dilation of vessels with oedema (swelling), lowered blood pressure and release of inflammatory cytokines. Normally the production of bradykinin is carefully balanced in the body. Some people have a tendency to release bradykinin. This results in spontaneous swelling - it is called hereditary episodic angioedema (HAE). There has been a treatment for HAE which has been in use since 2008. It is a medication called Icatibant. This blocks the effect of bradykinin at one of its receptors. It is given by injection under the skin. It has a short half life of approximately 1.5 hours.

The primary aim of the study is to see if treatment with Icatibant will improve blood oxygen levels. COVID-19 patients attending hospital with early symptom onset and low oxygen levels will screened for inclusion in the trial. Patients will be randomly allocated into one of two groups. One group will be given the study drug, Icatibant. The other group will be given a placebo injection containing saline water. Patients and research investigators will be blinded to treatment allocation.

Prior to receiving Icatibant/placebo, patients will have baseline measurements carried out. Blood pressure, Mean arterial pressure, heart rate, oxygen saturations and Fraction of inspired oxygen (FiO2) measurement will be carried out. Patients will undergo an arterial blood gas test. Part of the blood taken will be used for the measurement of interleukin-6 (IL-6) and part will be stored for future use. Patients will also have a retinal photograph of both eyes to assess the retinal vessel size. These measurements will be repeated 3 hours after receiving Icatibant/placebo.

A blood sample will also be taken from a group of control participants who do not have COVID-19 infection. The control blood samples will be analysed for IL-6 and part will also be stored for future use. The results will be compared to the baseline blood sample results taken from the COVID-19 positive trial patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Documented evidence of COVID-19 and symptom onset of 7 days or less
3. Acute hypoxia which will be defined as either low resting saturations <94% or supplementary oxygen to maintain oxygen saturations at >94%

Exclusion Criteria:

1. Patients known to be pregnant or breastfeeding.
2. Patients with unstable ischaemic heart disease or acute stroke
3. Patients enrolled in other clinical trials of an investigational medicine within the previous 28 day period
4. Patients who refuse to have blood samples taken.
5. Known hypersensitivity to Icatibant
6. Patients who at time of consent are likely to require imminent non-invasive/ invasive ventilatory support or patients already established on continuous positive airway pressure (CPAP).
7. Patients with chronic heart or lung disease whose oxygen levels are reduced, but are unchanged from baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change in Oxygenation | Baseline and 3 hours after study drug administration
  Alveolar-arterial gradient (Arterial blood gas sampling and FIO2 measurement)

SECONDARY OUTCOMES:
Change in Blood pressure | Baseline and 3 hours after study drug administration
  Systolic and diastolic blood pressure (mmHg)
Change in mean arterial pressure (MAP) | Baseline and 3 hours after study drug administration
  Measurement of mean arterial pressure (mmHg)
Change in heart rate | Baseline and 3 hours after study drug administration
  Measurement of pulse (beats/minute)

OTHER OUTCOMES:
Change in interleukin-6 levels | Baseline and 3 hours after study drug administration
  Blood sample will be taken for measurement of serum IL-6 (pg/ml)
Change in retinal vessel size (As measured by optical coherence tomography) | Baseline and 3 hours after study drug administration
  OCT retinal imaging of both eyes. Retinal vasculature will be assessed.
Oxygen requirements and saturations 24 hours post study drug | Approximately 24 hours after study drug administration
  Documentation of oxygen required and oxygen saturations

CONTACTS AND LOCATIONS:
Overall Officials: Joe Kidney, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Mater Infirmorum Hospital, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailey M, Linden D, Earley O, Guo Parke H, McAuley DF, Peto T, Taggart C, Kidney J. Inhibition of bradykinin in SARS-CoV-2 infection: a randomised, double-blind trial of icatibant compared with placebo (ICASARS). BMJ Open. 2023 Nov 30;13(11):e074726. doi: 10.1136/bmjopen-2023-074726. PMID 38035747